CLINICAL TRIAL: NCT03298724
Title: Teachers and Parents as Partners During Middle School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0872; R324B160043 (Other Grant/Funding Number: US Dept of Education); A173000 (Other: UW Madison); EDUC\EDUC PSYCHOLOGY (Other: UW Madison)
Record Dates: First submitted 2017-09-14; First posted 2017-10-02 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-04

CONDITIONS: Behavior Problem
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Single case experimental design (multiple baseline across setting)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAPP Intervention (Experimental): The Teachers and Partners intervention will be provided
  Interventions: Behavioral: Teachers and Parents as Partners

INTERVENTIONS:
Behavioral: Teachers and Parents as Partners — A family-school partnership intervention to improve the home-school connection, parenting and teaching strategies, and child behavior outcomes.
  Other Names: Conjoint Behavioral Consultation

SUMMARY:
There are two aims of this study (a) to examine the effect of Teachers and Parents as Partners on student, parent, and teacher outcomes in middle school and (b) identify barriers and facilitators to implementing Teachers and Parents as Partners in middle school for students with behavior concerns.

DETAILED DESCRIPTION:
Teachers and Parents as Partners will occur in a series of stages comprised of approximately four structured meetings over approximately 8 weeks. A Teachers and Parents as Partners consultant will meet together with a student's parent(s), teachers, other school personnel (as appropriate), and the student (as appropriate). The Teachers and Parents as Partners team will collaboratively address behavior problem solving objectives. Specific CBC objectives include: identifying strengths and specific behaviors of concern, specifying alternative prosocial behaviors, creating measurable behavior goals, co-constructing behavior intervention/support plans to address the target concerns, creating sustainable conditions to support plan implementation at home and school, and evaluating the plan to assess progress toward goals.

Treatment integrity in multiple dimensions (e.g., engagement, dosage, adherence) will be assessed at the two tiers of implementation (i.e., Teachers and Parents as Partners procedural integrity and behavior support plan implementation) to determine the extent to which procedures are implemented as designed.

During each structured meeting, Teachers and Parents as Partners consultants will inquire with parents, teachers, other school personnel, and students about barriers and facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Students will be eligible if they have scores in the "elevated" or "extremely elevated" risk categories on the parent and teacher version of the Behavior Assessment Scale for Children (BASC) 3 Behavioral and Emotional Screening System (BESS). Parents, and primary teachers and school staff associated with an eligible student will be included.

Exclusion Criteria:

* Students who do not meet the inclusion criteria will be excluded from participation, which includes their parent(s), teachers, and other school personnel. Students also may not be eligible if they have mental health concerns that may not be appropriate for Teachers and Parents as Partners or a research project (e.g., some internalizing problems, students who pose an risk of harming themselves).

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Direct Behavior Ratings (change over time) | up to 32 weeks
  Parents and teachers provide ratings of child behavior

OTHER OUTCOMES:
Teacher report of student work completion (change over time) | up to 32 weeks
  Teacher reported student work completion
Monitoring Scale (change over time) | up to 32 weeks
  Parent Monitoring Knowledge of child activities
Problem solving competencies | up to 32 weeks
  Parent and teacher reported problem solving competencies
Parent-teacher relationship scale (change over time) | up to 32 weeks
  Parents and teacher report on the parent-teacher relationship
Behavior Intervention Rating Scale Revised | up to 32 weeks
  Parent, teacher, and student satisfaction with procedures

CONTACTS AND LOCATIONS:
Overall Officials: Andy Garbacz, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided